CLINICAL TRIAL: NCT00223379
Title: Longitudinal Endodontic Study of Apical Preparation Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kenneth Hargreaves, Chair, Dept. of Endodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012-1904-342
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Apical Periodontitis of Pulpal Origin
Keywords: Apical Periodontitis, Root Canal Therapy, Apical Preparation
MeSH Terms: conditions — Periapical Periodontitis | interventions — Endodontics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endodontic procedure with varied apical preparation size — Comparison of two commonly used techniques for performing root canal treatment: 1) Lightspeed method 2)Buchannan method

SUMMARY:
This protocol is for a clinical trial evaluating the clinical success of root canal therapy performed on teeth with chronic apical periodontitis of pulpal origin with either large or small apical root canal preparation techniques.

DETAILED DESCRIPTION:
This randomized clinical trial will compare the clinical success of two commonly used techniques for performing non-surgical endodontic procedures on teeth with chronic apical periodontitis of pulpal origin. The first method, termed the "GT method" uses a commercially available rotary file system to instrument the root canal systems from the crown to the apical portion of the root. After completion of this technique, the apical portion of the root is prepared to the same standardized ISO size #20 in all roots (i.e., 0.2 mm cross-sectional diameter). The second method, termed the "Lightspeed method" uses a different commercially available rotary file system to shape the root canal systems from the apical to the crown portion of the root. After completion of this technique, the apical preparation is often larger in cross-sectional diameter than that observed after the GT method; however, an equally important distinction is that the Lightspeed method customizes the final cross-sectional diameter for each root canal system, and thus each root has a similar enlargement of apical preparation size due to proportionate removal of infected dentin at the end of the root. Although the Lightspeed method may result in reduced bacteria in the apical portion of root canal systems, there is no evidence to date that this effect improves clinical success rates. This study will test the hypothesis that the larger apical preparation size produced by the Lightspeed instrumentation system will produce a higher percentage of clinically successful treatments of teeth with apical periodontitis (AP) as compared to the GT method

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age.
2. Clinical indication for Non-Surgical Root Canal Therapy (NSRCT).
3. 1st or 2nd maxillary or mandibular molar.
4. Diagnosis must be Chronic Apical Periodontitis (CAP) with or without symptoms.
5. Intact, mature apices.
6. ASA I or II.

Exclusion Criteria:

1. Failure to meet any of the above
2. Previous NSRCT
3. Previous pulpotomy or pulpectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Radiographic and clinical evidence of osseous healing of chronic apical periodontitis of pulpal origin. | 2 year

SECONDARY OUTCOMES:
Pain | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karl Keiser, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio, Texas
Locations (1):
- The University of Texas Health Science Center, San Antonio, Texas, United States